CLINICAL TRIAL: NCT04796285
Title: A Validation Study of the Lab Clasp Device: A Point of Care Sepsis Risk Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Cambridge Medical Technologies, LLC (Industry)
Responsible Party: Principal Investigator, Guruprasad Jambaulikar, MBBS, MPH, Director of Research, Emergency Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P004159
Record Dates: First submitted 2021-02-26; First posted 2021-03-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sepsis; Sepsis Bacterial; Lactate Blood Increase; Infectious Disease
Keywords: point of care; sepsis; interstitial fluid; lactate
MeSH Terms: conditions — Sepsis; Hyperlactatemia; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Lab Clasp (Experimental): A finger based device to assay interstitial fluid lactate
  Interventions: Device: Lab Clasp

INTERVENTIONS:
Device: Lab Clasp — Finger-based interstitial fluid assessment device

SUMMARY:
The overall purpose of this study is to demonstrate the usability of a clinical-grade device in the form of a finger clasp similar to a pulse oximeter for monitoring lactate values, by comparing its performance in reading interstitial fluid lactate values against a known clinical standard in the form of venous lactate levels.

Serum lactate measurements are used clinically as a measure of end-organ dysfunction and physiologic stress. Changes in lactate may indicate worsening infection in the setting of sepsis, drug toxicity for certain xenobiotics, or exercise tolerance in exercise physiology. Serum lactate cutoffs have been developed for various disease states and trigger a variety of medical decisions directed at managing the course of the disease.

A common theme in the application of lactate measurements to understanding changes in physiology is the need to obtain venous blood to determine lactate. While point-of-care assays have been developed that improve the processing speed, there continues to be a need to obtain fingerstick blood or in most cases, venous blood. Obtaining venous blood for serum lactate requires an individual with phlebotomy skills, the processing capabilities of a laboratory to determine lactate concentrations, or the availability of point of care technology.

An alternative method to measure lactate is to sample interstitial fluid which surrounds cells and tissues in the body. Obtaining interstitial fluid is potentially less invasive without the need for repeat phlebotomy or the presence of an indwelling intravenous catheter which can become complicated by infection. The analysis of interstitial fluid for glucose has been validated and is clinically utilized in continuous glucose monitors in individuals with diabetes. In this investigation, the investigators will utilize a novel device, the Lab Clasp to obtain interstitial fluid in a noninvasive method. The Lab Clasp is manufactured to resemble a finger pulse oximeter with additional onboard microfluidics channels that obtain a lactate concentration from interstitial fluid. This streamlined process of obtaining the point of care lactate measurements on demand allows for tasks like serial lactate measurements to be accomplished on a reliable schedule with less workload for nursing staff typically required to draw venous blood. Additionally, the portable and noninvasive nature of the Lab Clasp system may render it usable in facilities that lack skilled staff necessary to perform phlebotomy.

ELIGIBILITY:
Inclusion Criteria

1. Are 18 years or older
2. In general good health, evidenced by no unstable medical problems (no medication changes in the past 3 months)
3. Have no known skin allergy to the components of the Lab Clasp
4. Willing to comply with all study procedures including providing venous blood samples at the CCI
5. Are English speaking
6. Provide consent to participate in the study

Exclusion Criteria:

1. Individuals <18 years old
2. General frailty of health
3. Prohibitively poor vascular access
4. History of malignancy or active malignancy
5. History of cardiac illness
6. History of HIV on antiretrovirals
7. History of alcohol abuse
8. History of uncontrolled psychiatric illness
9. Recent hospitalization within the past 30 days
10. History of vaping, propylene glycol use
11. History of statin use
12. Non-English speaking
13. Pregnant women, children, vulnerable populations
14. Investigator discretion for suspicion of poor study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of average difference lactate readings between Lab Clasp and laboratory reference values. | 150 minutes
  The primary outcome measure will be the average difference in lactate values between the Lab Clasp device and the reference (laboratory venous lactate) in healthy volunteers. We will obtain multiple (nine timepoints in total) investigational-reference measurement pairs in each subject (150 minutes total) and will average the difference over all pairs from all subjects.

SECONDARY OUTCOMES:
Measurement of participant experience | 150 minutes
  We will give each participant a questionnaire when they finish their visit and will ask for their experience (Likert-type scale, 1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Guruprasad Jambaulikar, MBBS, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No